CLINICAL TRIAL: NCT00208000
Title: A Clinical Double Blind, Randomized Study of the Efficacy of Hyperuricemia Treatment With Anserine Product.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMR93-IRB-22
Record Dates: First submitted 2005-09-16; First posted 2005-09-21 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2005-09

CONDITIONS: "Hyperuricemia,Anserine"
MeSH Terms: conditions — Hyperuricemia

INTERVENTIONS:
Drug: Marine active

SUMMARY:
Hyperuricemia is a common metabolic disorder.The Yaizu Suisankagaku Industry Company have developed industrial production named Marine Active, was able to offer anti-fatigue activity by animal trial data. Human clinical trials showed reduced creatine phosphokinase activity and a sero-uric acid reduction activity was also observed. So we are committed to design the clinical randomized, double blind study about hyperuricemia management with Marine Active. All these efforts are hoped to find a novel method to manage hyperuricemia.

DETAILED DESCRIPTION:
Hyperuricemia is a common metabolic disorder. It can result from a decreased renal uric acid excretion, increased urate production, or both. The classical association with clinical gout is well-known. The principal indications for uric acid-lowering therapy, including allopurinol, probenecid and sulfinpyrazone, are the patients with gout history, macroscopic subcutaneous tophi, frequent attacks of gouty arthritis, or a documented state of uric acid overproduction. Hyperuricemia without gout attack is not an indication for treatment.However, hyperuricemia is often associated with other cardiovascular disease risk factors such as obese, hyperlipidemia, glucose intolerance and hypertension. It is known a symptom of syndrome X (also known as multiple risk factor clustering syndrome). Diet control is the only way to control serum uric acid level, but always it is not enough. So how to management hyperuricemia is important and is a potential management.Histidine-containing dipeptides such as Anserine and Carnosine have been studied extensively in recent years. These dipeptides were shown to be effective in acting as buffering agents against protons developed during anaerobic exercise. Anserine and Carnosine also have strong anti-oxidant activity, anti-cancer activity, immuno-response modulation, fat reduction and enhanced wound healing functions. The Yaizu Suisankagaku Industry Company have developed industrial production process to extract and purify the dipeptides from Bonito and Tuna. The extract, named Marine Active, was able to offer anti-fatigue activity by animal trial data. Human clinical trials showed reduced creatine phosphokinase activity and a sero-uric acid reduction activity was also observed. So we are committed to design the clinical randomized, double blind study about hyperuricemia management with Marine Active. All these efforts are hoped to find a novel method to manage hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age between 18 to 60 years
* With the data of serum uric acid level more than 8.0 mg/dl within 2 weeks before the initiation of study
* Signed informed consent obtained prior to inclusion into the study

Exclusion Criteria:

* Pregnant women.
* Acute onset of gouty arthritis or renal stone
* Significant liver or renal dysfunction, hematological disease, oncological disease, or other life threatens disorders.
* Condition that need the management of diuretics or analgesics agent
* Have been administrated by anti-hyperuricemia agent or healthy food with in 4 weeks before the initiation of study.
* The serum uric acid level could be decrease to lower than 8 mg/dl by diet control.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2004-07; Study Completion 2006-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chiu-Shong Liu, Director, Principal Investigator — Family Medicine, China Medical University Hospital
Locations (1):
- China Medical University Hospita, Taichung, Taiwan